CLINICAL TRIAL: NCT03546478
Title: 99mTc Labelled Affibody SPECT/CT Imaging for Breast Cancer HER2 Characterization
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CaiJ
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: SPECT/CT; HER2 imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-ABH2 SPECT/CT (Experimental): The patients were injected with 370±54 MBq of 99mTc-ABH2 in one dose intravenously and underwent SPECT/CT scan 90-270 min later.
  Interventions: Biological: 99mTc-ABH2

INTERVENTIONS:
Biological: 99mTc-ABH2 — 99mTc-ABH2 were injected into the patients before the SPECT/CT scans
  Other Names: 99mTc labelled HER2 affibody

SUMMARY:
This is an open-label single photon emission tomography/computed tomography (SPECT/CT) study to investigate the diagnostic performance and evaluation efficacy of 99mTc-ABH2 in breast cancer patients. A single dose of 370±54 Mega-Becquerel (MBq)99mTc-ABH2 will be injected intravenously. Visual and semiquantitative method will be used to assess the SPECT/CT images.

DETAILED DESCRIPTION:
99mTc-ABH2 is an affibody probe targeting HER2. The investigators will determine the use of 99mTc-ABH2 SPECT/CT in the detection of HER2-positive breast cancer, and to compare its diagnostic value with routine immunohistochemistry (IHC) pathological staining. HER2 imaging, specifically to HER2 receptor expressed on malignant breast cancer cell surface, might help for targeted therapy with monoclonal antibody such as trastuzumab in breast cancer, and may improve the treatment strategy of breast cancer. The investigator will determine the use of 99mTc-ABH2 SPECT/CT in stratifying breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients with breast cancer before surgery Conventional imaging within 1 month Signed written consent Age above 29 years Female

Exclusion Criteria:

Pregnancy Breastfeeding Renal function: serum creatinine > 3.0 mg/dl Known allergy against affibody Any medical condition that, in the opinion of the investigator, may significantly interfere with study compliance

Ages: 29 Years to 76 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
T/B | 1 year
  Target/Background ratio of 99mTc-ABH2 SPECT/CT in Diagnosis of HER2-positive breast cancer

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical Colleg
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China